CLINICAL TRIAL: NCT03641365
Title: Accuracy of Computer-assisted Template-based Implant Placement Using CAD/CAM Stereolithographic Surgical Templates With or Without Metallic Sleeves: a Randomized Controlled Trial
Brief Title: Sleeves Versus Sleeveless Template
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osstem AIC (Other)
Responsible Party: Principal Investigator, Marco Tallarico, Principal Investigator, Osstem AIC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Osstem_001
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Guided Surgery Accuracy; Dental Implant Failed; Complications
Keywords: Intraoral scanner; Guided surgery; Implant accuracy; Dental implants
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of parallel group design conducted at one centre.
Who Masked: Outcomes Assessor
Masking Description: An expert blinded mechanical engineer (FC) performed all the measurements. Post-operative STL files were sent with a code, without indicating patient's group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Test group: Surgical template without metallic sleeves. In this case the surgical template has all been designed and fabricated in acrylic material by mean of stereolitographic technology.
  Interventions: Device: Test group
- Control group (Active Comparator): Control group: Surgical template with metallic sleeves. Surgical template has designed and fabricated in acrylic material by mean of stereolitographic technology and metallic sleeves have been bonded after its production.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Test group — Guided Implant placement Positioning/placement of dental implants thought the fully acrylic surgical template without metallic sleeves.
  Other Names: Sleeveless Template
  Arms: Test group
Device: Control group — Guided Implant placement Positioning/placement of dental implants thought the acrylic surgical template with metallic sleeves.
  Other Names: Conventional Template
  Arms: Control group

SUMMARY:
To compare virtual planning accuracy of computer-assisted template-based implant placement using CAD/CAM stereolithographic surgical templates with or without metallic sleeves.Furthermore to compare open versus closed holes in case of sleeveless templates.

Any partially edentulous patients requiring at least one implant to be planed according to a computer-assisted template-based protocol were enrolled. Patients were randomised according to a parallel group design into two arms: surgical template with or without metallic sleeves. Three deviation parameters (angular, horizontal, vertical) were defined to evaluate the discrepancy between the planned and placed implant positions.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial of parallel group design conducted at one centre, between May 2016 and March 2017. The study was performed after approval was received from the institutional review board of the Aldent University, Tirana, Albania (2/2017).

The investigation was conducted according to the principles embodied in the Helsinki Declaration of 1975 for biomedical research involving human subjects, as revised in 2013. All patients were informed about the nature of the treatment and their written consent was obtained. Data collection was designed to preserve patient anonymity.

- Inclusion/exclusion criteria:

Any partially edentulous patient, aged 18 years or older, able to sign an informed consent, in need of an implant-supported fixed restoration was considered eligible for this study. Any potential implant location based on individual patient requirements was considered eligible in the present trial. Patients were not admitted to the study if any of the following exclusion criteria was present: general medical contraindication to oral surgery (American Society of Anesthesiologist, ASA, class III or IV); irradiation in the head and neck area less than one year before implantation; psychiatric problems; alcohol or drug abuse; pregnant or nursing; untreated periodontitis; severe bruxism or clenching; uncontrolled diabetes; poor oral hygiene and motivation; and inability to complete the follow-up.

Enrolled patients received preoperative photographs, periapical radiographs or panoramic x-rays for initial screening and evaluation. The prosthetic-driven planning workflow started by taking a cone beam computed tomography (CBCT) scan (Cranex 3Dx, Soredex, Tuusula, Finland) by using a wax bite to separate dental arches. Then, the patients received intraoral digital impression taken using the 3M True Definition Scanner (3M Italia, Pioltello, Milano). The digital data (STL, STereo Lithography interface format) was imported in a 3D design software (exocad DentalCAD, Exocad GmbH, Darmstadt, Germany) to realize a virtual wax-up according to the functional and esthetic requirements. Then, the STL and DICOM (Digital Imaging and COmmunications in Medicine) data were imported in a 3D software planning program (3Diagnosys ver. 5.0, 3DIEMME srl, Cantù, Italy). Then, the reprocessed surface extrapolated from the DICOM data (by using a Hounsfield scale filter) and the surface generated by the master cast scanning process, or by the intraoral scanning process, were merged with the best-fitting repositioning tools of the software (3Diagnosys ver. 5.0, 3DIEMME srl). At this point, prosthetic-driven implants/abutments size and location were planned taking into account the bone quality and quantity, soft tissue thickness, anatomical landmarks, as well as, type, volume and shape of the final restoration. After careful functional and esthetic evaluation and final verification, the prosthetic-driven plan was approved. At this point, patients were randomly assigned to receive conventional stereolithographic surgical template with (control group) or without (test group) metallic sleeves. Stereolithographic surgical templates were designed and fabricated by an independent certified center not previously involved in the study (New Ancorvis srl, Bargellino, Italy). In the test group, conventional templates with close-sleeve-design were produced to place implants between premolars. In case of implants to be place in molar area, template with open sites were produced to solve intermaxillary space limits.

- Surgical protocol:

One hour before implant placement, all patients underwent professional oral hygiene, prophylactic antiseptic with 0.2% chlorhexidine (Curasept, Curaden Healthcare, Saronno, Italy) for one minute, and prophylactic antibiotic therapy (2 g of amoxicillin or clindamycin 600 mg if allergic to penicillin). The fit of the surgical templates were accurately tried in the patient mouth to achieve a stable fit (Fit Checker, GC - Tokyo, Japan). All patients were treated under local anesthesia using articaine with adrenaline 1:100000 administered 20 minute before surgery. The surgical templates were stabilized on the residual teeth and fixed with two to three preplanned anchor pins.Hopeless teeth were extracted at the end of the intervention in order to improve the stability of the surgical template and to provide more reference point for measurements of the implant accuracy. Nevertheless, in case of immediate postextractive implants, residual teeth were extracted as atraumatically as possible immediately before surgery. In the test group, planned implants (Osstem TSIII, Osstem, Seoul, South Korea) were placed flapless using dedicate drills (OneGuide Kit, Osstem) in combination with a sleeveless surgical guide. In this case the drills were used directly thought the sleeve-designed template without metallic tubs and with not the need of drill reductions. In the control group, planned implants (Osstem TSIII, Osstem, Seoul, South Korea) were placed flapless using dedicate drills (OsstemGuide Kit[Taper], Osstem) in combination with reduction tools, within the surgical templates containing metallic sleeves. If the keratinized gingiva and the amount of bone were adequate, the implants were placed flapless. Otherwise, a flap was elevated and then the wound was closed with single-stitch sutures using 4.0 resorbable suture material (Vicryl, Ethicon J&J International, Sint-Stevens-Woluwe, Belgium). Implant site were prepared based on the bone density evaluated by the surgeon at the first drill. All the implant were inserted according to a one-stage protocol, with an insertion torque ranging from 35 to 45 Ncm. In case of poor bone density, the implant site was underprepared. Immediately after implant placement, patients of both groups receive a digital impression (3M True Definition Scanner, 3M Italia, Pioltello, Milano) taken at implant level using a dedicate abutments (Scan body type AQ, New Ancorvis srl), to check the position of the placed implants.

Following implant placement, all patients received oral and written recommendations about medication, oral hygiene maintenance and diet. Implants were loaded after 8 to 12 weeks of healing. Then, patients were followed twice a year for hygiene maintenance and occlusal control.

* Outcome measurements:

  * Implant failure: an implant was considered to be a failure if it was lost for mobility, implant fracture and/or any infection dictating implant removal. The stability of each individual implant was measured manually with a torque of 20 Ncm at delivery of the final restoration and later, with the prosthesis removed, if needed (infection, extensive peri-apical bone loss, mucosal inflammation).
  * Template-related complications: early surgical complications involved the surgical template comprised limited access in posterior areas, buccal bony dehiscence (due to a mismatching of the surgical template) evaluated sounding the implant site with a periodontal probe (PCPUNC156, Hu-Friedy Italy, Milan, Italy) before implant placement, insertion of different implant than planned, and fracture of surgical template. All the complications were recorded during follow-up by the same clinician (Marco Tallarico), who performed all the surgical procedures.
  * Accuracy: Three deviation parameters (horizontal, vertical, and angular) were defined and calculated between the planned and placed implant positions. The post-operative STL file, derived from the intraoral scan, was geometrically aligned with the files exported from the planning, by automated image registration using maximization of mutual information (Dental SCAN, ver.6, Open Technologies srl, Brescia, Italy). The horizontal (lateral), vertical (depth) and angular deviation between virtual and placed implants were calculated along the long axis of each implants. An expert blinded mechanical engineer (FC) performed all the measurements.
* Randomization:

One computer-generated restricted randomization list was created. Only one of the investigators, not involved in the selection and treatment of the patients, was aware of the random sequence and could have access to the randomization lists stored in a password-protected portable computer. The random codes were enclosed in sequentially numbered, identical, opaque, sealed envelopes. Envelopes were opened sequentially after the prosthetic-driven plan was approved.

- Statistical analysis:

Patient data were collected in a Numbers spreadsheet (Version 3.6.1 for Mac OS X 10.11.4). A bio-statistician with expertise in dentistry analyzed the data using SPSS software for Mac OS X (version 22.0; SPSS Inc., Chicago, IL, USA) for statistical analysis. Descriptive analysis was performed for numeric parameters using mean±standard deviation and median with confidence interval (95% CI). Implant failure and template-related complications between the two groups were compared using Fisher's exact probability test. The mean differences of the overall deviation in the clinical outcomes compared to the virtual plan, were compared between groups using a mixed-model repeated-measures analysis of variance (ANOVA). In the sleeve-less group, accuracy of open versus closed holes were also evaluated. All statistical comparisons were conducted with a P value set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patient
* Aged 18 years or older
* Able to sign an informed consent
* In need of an implant-supported fixed restoration

Exclusion Criteria:

* General medical contraindication to oral surgery (American Society of Anesthesiologist, ASA, class III or IV) including uncontrolled diabetes
* Irradiation in the head and neck area less than one year before implantation
* Psychiatric problems
* Alcohol or drug abuse
* Pregnant or nursing
* Untreated periodontitis or poor oral hygiene and motivation
* Severe bruxism or clenching
* Inability to complete the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Accuracy (discrepancy between virtual implant planning and placed implants) | Implant placement (baseline)
  Three deviation parameters (horizontal, vertical, and angular) were defined and calculated between the planned and placed implant positions. The post-operative STL file, derived from the intraoral scan, was geometrically aligned with the files exported from the planning, by automated image registration using maximization of mutual information (Dental SCAN, ver.6, Open Technologies srl, Brescia, Italy). The horizontal (lateral), vertical (depth) and angular deviation between virtual and placed implants were calculated along the long axis of each implants. An expert blinded mechanical engineer (FC) performed all the measurements.

SECONDARY OUTCOMES:
Implant failure | 4 months after implant placement (baseline)
  An implant was considered to be a failure if it was lost for mobility, implant fracture and/or any infection dictating implant removal. The stability of each individual implant was measured manually with a torque of 20 Ncm at delivery of the final restoration and later, with the prosthesis removed, if needed (infection, extensive peri-apical bone loss, mucosal inflammation).
Template-related complications | Implant placement
  Early surgical complications involved the surgical template comprised limited access in posterior areas, buccal bony dehiscence (due to a mismatching of the surgical template) evaluated sounding the implant site with a periodontal probe (PCPUNC156, Hu-Friedy Italy, Milan, Italy) before implant placement, insertion of different implant than planned, and fracture of surgical template.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tallarico, Dr, Principal Investigator — Studio Marco Tallarico
Locations (1):
- Studio Odontoiatrico Marco Tallarico, Rome, Italy

REFERENCES:
- [Background] D'haese J, Van De Velde T, Elaut L, De Bruyn H. A prospective study on the accuracy of mucosally supported stereolithographic surgical guides in fully edentulous maxillae. Clin Implant Dent Relat Res. 2012 Apr;14(2):293-303. doi: 10.1111/j.1708-8208.2009.00255.x. Epub 2009 Nov 10. PMID 19906267
- [Background] D'haese J, Ackhurst J, Wismeijer D, De Bruyn H, Tahmaseb A. Current state of the art of computer-guided implant surgery. Periodontol 2000. 2017 Feb;73(1):121-133. doi: 10.1111/prd.12175. PMID 28000275
- [Background] Tallarico M, Esposito M, Xhanari E, Caneva M, Meloni SM. Computer-guided vs freehand placement of immediately loaded dental implants: 5-year postloading results of a randomised controlled trial. Eur J Oral Implantol. 2018;11(2):203-213. PMID 29806667

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03641365/SAP_000.pdf